CLINICAL TRIAL: NCT03485365
Title: A Two-part Phase I Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics and Target Engagement of Single Intravenous and Subcutaneous Doses of GSK3858279 in Healthy Participants and to Evaluate the Efficacy of Repeat Subcutaneous Doses in Participants With Osteoarthritis of the Knee
Brief Title: A Safety, Tolerability, Pharmacokinetics (PK) and Target Engagement (TE) Study of GSK3858279 in Healthy Participants and Evaluation of the Efficacy of Repeat Doses in Participants With Osteoarthritis (OA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 207804; 2017-004809-41 (EudraCT Number)
Record Dates: First submitted 2018-03-27; First posted 2018-04-02 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Pain, Inflammatory
Keywords: Pain; Osteoarthritis of the knee; Target engagement; GSK3858279; Pharmacokinetics; Sequential
MeSH Terms: conditions — Pain; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in 3:1 ratio to receive GSK3858279 and placebo in sequential manner in Part A. In Part B, participants will be randomized in parallel groups to receive either GSK3858279 or placebo.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study. Participant and investigator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part A: Cohort 1: GSK3858279 (Experimental): Eligible participants will receive GSK3858279 via IV route.
  Interventions: Drug: GSK3858279 IV
- Part A: Cohort 2: GSK3858279 (Experimental): Eligible participants will receive GSK3858279 via IV route.
  Interventions: Drug: GSK3858279 IV
- Part A: Cohort 3: GSK3858279 (Experimental): Eligible participants will receive GSK3858279 via IV route.
  Interventions: Drug: GSK3858279 IV
- Part A: Cohort 4: GSK3858279 (Experimental): Eligible participants will receive GSK3858279 via IV route.
  Interventions: Drug: GSK3858279 IV
- Part A: Cohort 5: GSK3858279 (Experimental): Eligible participants will receive GSK3858279 via IV route.
  Interventions: Drug: GSK3858279 IV
- Part A: Cohort 6: GSK3858279 (Experimental): Eligible participants will receive GSK3858279 via SC route.
  Interventions: Drug: GSK3858279 SC
- Part A: Placebo (Placebo Comparator): Eligible participants will receive placebo matching to GSK3858279 via SC or IV route.
  Interventions: Drug: Placebo matching to GSK3858279 (SC or IV)
- Part B: GSK3858279 (Experimental): Eligible participants will receive GSK3858279 via SC route.
  Interventions: Drug: GSK3858279 SC
- Part B: Placebo (Placebo Comparator): Eligible participants will receive placebo matching to GSK3858279 via SC route.
  Interventions: Drug: Placebo matching to GSK3858279 (SC)

INTERVENTIONS:
Drug: GSK3858279 IV — GSK3858279 will be available as solution for injection to be administered via IV route.
  Arms: Part A: Cohort 1: GSK3858279; Part A: Cohort 2: GSK3858279; Part A: Cohort 3: GSK3858279; Part A: Cohort 4: GSK3858279; Part A: Cohort 5: GSK3858279
Drug: GSK3858279 SC — GSK3858279 will be available as solution for injection to be administered via SC route.
  Arms: Part A: Cohort 6: GSK3858279; Part B: GSK3858279
Drug: Placebo matching to GSK3858279 (SC or IV) — Placebo will be available as sodium chloride solution to be administered via SC or IV route.
  Arms: Part A: Placebo
Drug: Placebo matching to GSK3858279 (SC) — Placebo will be available as sodium chloride solution to be administered via SC route.
  Arms: Part B: Placebo

SUMMARY:
This study is the first administration of GSK3858279 in humans and will be conducted in two parts: Part A will consist of a single ascending dose escalation design to evaluate safety, tolerability, PK, TE and immunogenicity of either a single intravenous (IV) or a single subcutaneous (SC) dose. Approximately 48 healthy participants will be enrolled in 6 cohorts and randomized to 3:1 ratio (GSK3858279 or placebo). Part B will evaluate safety, tolerability, efficacy (pain), PK, TE and immunogenicity after repeat SC dosing. Approximately 50 OA participants will be randomized in a parallel group design to receive either GSK3858279 or placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

For Part A:

* Participants between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Volunteers who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body weight within the range 50 to 100 kilogram (kg) and body mass index (BMI) within the range 18 to 32 kilogram per meter square (kg/m^2) (inclusive).
* Male participants are eligible to participate if they agree to the following for at least 28 weeks after the dose of study intervention: Refrain from donating sperm PLUS either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR must agree to use contraception/barrier as detailed below: agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
* A female participant is eligible to participate if she is of non-reproductive potential.
* Capable of giving signed informed consent.

For Part B:

* Age between 40 and 75 years of age inclusive, at the time of signing the informed consent.
* OA of the index knee as defined by symptomatic for >=6 months with a clinical diagnosis of OA as per American College of Rheumatology (ACR) clinical diagnosis criteria.
* Average of daily pain score >=4 and <=9 by 11 point NRS (0 to 10) in index knee over 7 days prior to dosing (Day-7 to Day-1). Data should be recorded on at least 5 of 7 occasions by the participant to obtain a valid Baseline value.
* Kellgren and Lawrence (KL) score >=2 on X-ray obtained during screening. In addition, for participants with bilateral Knee OA, the index knee is determined at Baseline as the participant reported most painful knee over the 4 weeks prior to Baseline.
* A history of insufficient pain relief from, or inability to tolerate, or contraindication to, oral Non-steroidal anti-inflammatory drugs (NSAIDs).
* A participant must be willing and able to understand and participate in all scheduled evaluations and to complete all required tests and procedures including the use of patient diaries. This will be judged by the Investigator during the screening period.
* BMI within the range 19-34.9 kg/m^2 (inclusive)
* Male participants are eligible to participate if they agree to the following for at least 28 weeks after the dose of study intervention: refrain from donating sperm PLUS either: Be abstinent from heterosexual or homosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or must agree to use contraception/barrier as detailed: Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
* A female participant is eligible to participate if she is of non-reproductive potential.
* Capable of giving signed informed consent.

Exclusion Criteria:

For Part A:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Personal or family history of cardiomyopathy.
* Abnormal blood pressure at screening as determined by the investigator.
* History of symptomatic herpes zoster.
* Evidence of active or latent tuberculosis (TB) as documented by medical history, examination, and TB testing with a positive (not indeterminate) QuantiFERON test.
* Significant allergies to humanized monoclonal antibodies as per principal investigator's and GlaxoSmithKline (GSK) medical monitor's judgments.
* History or evidence of clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Lymphoma, leukemia, or any malignancy except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Alanine transaminase (ALT) >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Corrected QT (QTc) >450 milliseconds (msec).
* History of Stevens Johnson Syndrome.
* Known immunodeficiency.
* Participants with a chronic infection (example given [e.g.], osteomyelitis), who have been receiving treatment within three months prior to dosing or individuals with an active infection.
* Previous or current history of bleeding diathesis.
* Previous history of hypertrophic or keloid scarring.
* Intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing until final follow-up visit.
* Live vaccine(s), or plans to receive such vaccines within 1 month of screening until final follow-up visit.
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Treatment with antiplatelet or anticoagulant agents within 7 days of dosing.
* Major surgery (as per investigator's judgment) within 3 months prior to dosing.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 3 months.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation in any other clinical study involving an investigational study intervention or any other type of medical research within the last 30 days, 5 half-lives or twice the duration of the biological product before dosing day in the current study.
* Presence of Hepatitis B surface antigen (HBsAg) at screening.
* Presence of the Hepatitis B core antibody (HBcAb) at screening.
* Positive Hepatitis C antibody test result at screening.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* Abnormal clinically significant echocardiogram at screening, as assessed by the investigator.
* Cardiac troponin levels out of normal range at screening.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of >21 units for males and >14 units for females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Smokelyser levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Regular use of known drugs of abuse.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

For Part B:

* Diagnosis of one or more of the following, as per medical records: Significant pain in any joint other than the index knee or any referred pain that would impact ability to assess pain in the index knee as per investigator's judgement (Pain in other locations should be less than pain in target knee).
* Current inflammatory arthritis such as rheumatoid arthritis, autoimmune disorder affecting joints, seronegative spondyloarthritis, gout or pseudogout in any joint (defined as acute episodic attacks of swollen, painful joint in a participant with X-Ray chondrocalcinosis or calcium pyrophosphate dehydrate [CPPD] crystals).
* History of gout or pseudogout in any large joint.
* History or evidence of infectious arthritis, Paget's disease, ochronosis, Wilson's disease, primary osteochondromatosis, osteonecrosis and other causes of significant joint disease osteoarthritis as determined by the investigator.
* History of fibromyalgia.
* Current immunodeficiency diseases.
* Current osteoporosis with symptomatic vertebral or hip fractures.
* Current regional pain syndromes caused by lumbar or cervical compressions with radiculopathy.
* History of significant medical illness in the opinion of the investigator would interfere with the study procedures and / or assessments.
* Symptomatic herpes zoster within 3 months prior to screening.
* Evidence of active or latent TB as documented by medical history, examination and TB testing: either a positive tuberculin skin test (TST; defined as a skin induration >5 millimeter (mm) at 48 to 72 hours, regardless of Bacillus Calmette-Guerin (BCG) or other vaccination history) or a positive (not indeterminate) QuantiFERON test.
* History of significant allergies to humanized monoclonal antibodies.
* History or evidence of clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linearIgA dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis.
* History of malignancy within the last 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* ALT >1.5 times the ULN.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent)
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTc >450 msec or QTc >480 msec in participants with bundle branch block.
* History of primary cardiomyopathy and any major cardiac or vascular event within the last 6 months, including and not limited to myocardial infarction, unstable angina, cerebrovascular event, peripheral arterial or venous thrombosis.
* Current or history of renal disease, or estimated creatinine clearance <60 mL/minute/1.73/ m^2 or serum creatinine >1.5 times the ULN or urine albumin:creatine ratio of >300mg/g at screening.
* Planned surgical procedure over the duration of the study.
* Previous or current history of bleeding diathesis, excessive bleeding or coagulation disorders.
* History of Stevens Johnson Syndrome.
* Participants with active, recurrent or chronic infection (e.g., osteomyelitis), who have been receiving treatment within three months prior to dosing or individuals with an active infection.
* History of significant trauma or surgery to a knee, hip or shoulder within the last 6 months.
* Radiographic evidence of sub-chondral fractures or radiographic abnormalities not consistent with osteoarthritis of the index knee at screening.
* Live vaccine(s) within 1 month prior to screening, or plans to receive such vaccines during the study.
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Intra-articular therapy within 3 months prior to signing the informed consent.
* Immunosuppressant's, including corticosteroids (parenteral within 3 months of screening; oral within 1 month of screening).
* Unable or unwilling to discontinue all pain medication including topical analgesic or adjunctive treatment.
* Major surgery (as per investigator's judgement) within 3 months prior to dosing.
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within 56 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the dosing day.
* Current enrolment or past participation in a clinical study of an investigational drug intervention within the last 3 months or 5 half-lives (whichever is longer) of signing consent.
* Positive HIV antibody test.
* Presence of HBsAg at screening.
* Positive Hepatitis C antibody test result.
* Positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention.
* Positive coronavirus (Coronavirus Disease strain 19 [COVID-19]: Severe acute respiratory syndrome- Coronavirus-strain 2 [SARS-CoV-2] polymerase chain reaction [PCR] test of a combined throat and nasopharyngeal swab).
* Clinically significant abnormal ECG at screening, as assessed by the investigator.
* Cardiac troponin or N-terminal pro B-type natriuretic peptide (NT-proBNP) levels out of normal range at screening.
* A positive pre-study drug/alcohol screen at screening.
* Regular alcohol consumption within 6 months prior to signing the informed consent defined as: an average weekly intake of >14 units for males and >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Regular use of known drugs of abuse
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- GSK Investigational Site, Berlin, Germany
- GSK Investigational Site, Warsaw, Poland
- United Kingdom (3):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part study. Part A was a sequential group with a single ascending dose escalation in healthy participants. Single intravenous (IV) doses and a single subcutaneous (SC) dose were investigated in separate cohorts of participants. Part B was parallel group with repeat SC dosing of GSK3858279 or matching placebo in participants with Knee Osteoarthritis.
Pre-assignment Details: A total of 97 participants were enrolled in the study. Out of which 49 participants enrolled in Part A and 48 participants in Part B of the study.
Groups:
- Part A: Cohort 1: GSK3858279: Healthy participants received single doses of GSK3858279 0.1 mg/kg through IV route in Cohort 1. The participants were followed up for 84 days post dosing in Cohort 1.
- Part A: Cohort 2: GSK3858279: Healthy participants received single doses of GSK3858279 0.3 mg/kg through IV route in Cohort 2. The participants were followed up for 112 days post dosing in Cohort 2.
- Part A: Cohort 3: GSK3858279: Healthy participants received single doses of GSK3858279 1 mg/kg through IV route in Cohort 3. The participants were followed up for 112 days post dosing in Cohort 3.
- Part A: Cohort 4: GSK3858279: Healthy participants received single doses of GSK3858279 3 mg/kg through IV route in Cohort 4. The participants were followed up for 112 days post dosing in Cohort 4.
- Part A: Cohort 5: GSK3858279: Healthy participants received single doses of GSK3858279 10 mg/kg through IV route in Cohort 5. The participants were followed up for 140 days post dosing in Cohort 5.
- Part A: Cohort 6: GSK3858279: Healthy participants received single doses of GSK3858279 3 mg/kg through SC route in Cohort 6. The participants were followed up for 140 days post dosing in Cohort 6.
- Part A: Pooled Placebo: Healthy participants received single doses of matching Placebo to GSK3858279 through IV or SC route. The participants were followed up based on the treatment they received from 84 to 140 days post dosing.
- Part B: Cohort 7: GSK3858279: Participants with knee Osteoarthritis (OA) received weekly repeat doses of GSK3858279 240 mg through SC route up to day 56. The participants were followed up for 84 days post dosing in Cohort 7.
- Part B: Placebo: Participants with knee osteoarthritis received weekly repeat doses of placebo matching to GSK3858279 via SC route up to day 56. The participants were followed up for 84 days post dosing.
Period: Overall Study
Arm/Group | Part A: Cohort 1: GSK3858279 | Part A: Cohort 2: GSK3858279 | Part A: Cohort 3: GSK3858279 | Part A: Cohort 4: GSK3858279 | Part A: Cohort 5: GSK3858279 | Part A: Cohort 6: GSK3858279 | Part A: Pooled Placebo | Part B: Cohort 7: GSK3858279 | Part B: Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 24 | 24
Completed | 6 | 6 | 6 | 5 | 6 | 6 | 12 | 24 | 24
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1: GSK3858279 | Part A: Cohort 2: GSK3858279 | Part A: Cohort 3: GSK3858279 | Part A: Cohort 4: GSK3858279 | Part A: Cohort 5: GSK3858279 | Part A: Cohort 6: GSK3858279 | Part A: Pooled Placebo | Part B: Cohort 7: GSK3858279 | Part B: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 24 | 24 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 5 | 6 | 6 | 6 | 13 | 17 | 18 | 83
  >=65 years | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 7 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 8 | 13 | 27
  Male | 5 | 6 | 4 | 6 | 5 | 4 | 13 | 16 | 11 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 4
  BLACK OR AFRICAN AMERICAN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  WHITE | 6 | 5 | 6 | 4 | 5 | 6 | 13 | 23 | 24 | 92

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. TEAE is defined as an AE that occurred on or after the first dose date of study intervention. SAEs is defined as any serious adverse event that, at any dose which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, other situations as per investigator's medical or scientific judgment.
Time Frame: Up to 141 days
Population: Safety Population comprised of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: GSK3858279 | Part A: Cohort 2: GSK3858279 | Part A: Cohort 3: GSK3858279 | Part A: Cohort 4: GSK3858279 | Part A: Cohort 5: GSK3858279 | Part A: Cohort 6: GSK3858279 | Part A: Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 13
Participants
  Participants with TEAEs | 2 | 2 | 4 | 6 | 6 | 6 | 12
  Participants with SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. TEAE is defined as an AE that occurred on or after the first dose date of study intervention. SAEs is defined as any serious adverse event that, at any dose which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, other situations as per investigator's medical or scientific judgment.
Time Frame: Up to 141 days
Population: Safety Population comprised of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 7: GSK3858279 | Part B: Placebo
Number analyzed (Participants) | 24 | 24
Participants
  Participants with TEAEs | 21 | 15
  Participants with SAEs | 0 | 0

3. Primary Outcome: Part A: Number of Participants With Clinically Significant Changes in Hematology, Clinical Chemistry Laboratory Parameters and Urinalysis
Description: The parameters evaluated for Hematology were Basophils, Eosinophils, Hematocrit, Hemoglobin (Hg), Lymphocytes, mean corpuscular Hg, mean corpuscular volume, Monocytes, Platelet count, Red blood cells, Reticulocytes, Total Neutrophils, White blood cells count (WBC). For Clinical Chemistry- Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Bilirubin, Calcium, Creatinine, Direct bilirubin, Glucose, Potassium, Sodium, Total bilirubin, Total protein, TroponinT, N-terminal pro B-type natriuretic peptide (NT-ProBNP) and Urea. For Urinalysis-Urine bilirubin, Occult blood, Glucose, Ketones, Nitrates, pH, Protein, Specific gravity, Urobilinogen and Leukocyte Esterase for detecting WBC. Changes from baseline in hematology, clinical chemistry and urinalysis were reviewed by the investigator, medical monitor and safety physician to determine clinical significance; the number of participants with clinically significant changes is reported.
Time Frame: Up to 141 days
Population: Safety Population comprised of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: GSK3858279 | Part A: Cohort 2: GSK3858279 | Part A: Cohort 3: GSK3858279 | Part A: Cohort 4: GSK3858279 | Part A: Cohort 5: GSK3858279 | Part A: Cohort 6: GSK3858279 | Part A: Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 13
Participants
  Hematology | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinical Chemistry | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Hematology, Clinical Chemistry Laboratory Parameters and Urinalysis
Description: as for outcome 3
Time Frame: Up to 141 days
Population: Safety Population comprised of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 7: GSK3858279 | Part B: Placebo
Number analyzed (Participants) | 24 | 24
Participants
  Hematology | 0 | 0
  Clinical Chemistry | 0 | 0
  Urinalysis | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Clinically Significant Changes in Electrocardiogram Findings
Description: Twelve-lead Electrocardiogram (ECG) were performed in a semi-supine position using an ECG machine that automatically calculates the heart rate and measures PR interval, QRS duration, Uncorrected QT and corrected QT intervals (QTc) intervals. Changes from baseline in ECG findings were reviewed by the investigator, medical monitor and safety physician to determine clinical significance; the number of participants with clinically significant changes is reported.
Time Frame: Up to 141 days
Population: Safety Population comprised of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: GSK3858279 | Part A: Cohort 2: GSK3858279 | Part A: Cohort 3: GSK3858279 | Part A: Cohort 4: GSK3858279 | Part A: Cohort 5: GSK3858279 | Part A: Cohort 6: GSK3858279 | Part A: Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Electrocardiogram Findings
Description: as for outcome 5
Time Frame: Up to 141 days
Population: Safety Population comprised of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 7: GSK3858279 | Part B: Placebo
Number analyzed (Participants) | 24 | 24
Participants | 0 | 0

7. Primary Outcome: Part A: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs included systolic and diastolic blood pressure, pulse and respiratory rate and were measured with the participant in semi-supine position after 5 minutes rest. Temperature was also measured as a vital sign but did not require positioning or rest prior to measuring. Changes from baseline in vital signs were reviewed by the investigator, medical monitor and safety physician to determine clinical significance; the number of participants with clinically significant changes is reported.
Time Frame: Up to 141 days
Population: Safety Population comprised of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1: GSK3858279 | Part A: Cohort 2: GSK3858279 | Part A: Cohort 3: GSK3858279 | Part A: Cohort 4: GSK3858279 | Part A: Cohort 5: GSK3858279 | Part A: Cohort 6: GSK3858279 | Part A: Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Vital Signs
Description: as for outcome 7
Time Frame: Up to 141 days
Population: Safety Population comprised of all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 7: GSK3858279 | Part B: Placebo
Number analyzed (Participants) | 24 | 24
Participants | 0 | 0

9. Primary Outcome: Part B: Change From Baseline in Knee Pain as Assessed by Average of Daily Pain Numeric Rating Scale at Week 8
Description: Change from Baseline in knee pain due to Osteoarthritis were reported by average of daily pain numeric rating scale (NRS) at Week 8. The pain NRS is an 11-point scale (ranging from 0-10) for self-reporting of average knee pain where 0 indicates no pain, and 10 indicates the worst possible pain. For each participant, the mean pain score prior to each visit was calculated as the average pain intensity in the 7 days prior to assessment visit. Participants were instructed to complete the pain NRS questionnaire at approximately the same time each day. A negative value change from baseline indicates an improvement. Baseline scores for each participant were assigned based on the first dosing visit.
Time Frame: Baseline (Day 1) and Week 8
Population: Intent-to-Treat population comprised of all randomized participants who received at least one dose of study intervention. Two participants were randomized to Placebo and withdrew from study intervention post baseline due to adverse events; data following study intervention withdrawal were not included and outcomes for the analysis were assumed to be similar to participants who completed the study intervention.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part B: Cohort 7: GSK3858279 | Part B: Placebo
Number analyzed (Participants) | 24 | 22
Scores on a scale | -2.82 (1.752) | -1.62 (1.709)
Statistical Analysis 1: Comparison: Part B: Cohort 7: GSK3858279 vs Part B: Placebo; Test type: Other — Bayesian Repeated Measures Model; Median Difference (Net) = -1.18, 95% CI 2-sided [-2.15 to -0.20], Standard Deviation 0.494 — Posterior median difference (GSK3858279 - Placebo) and 95% credible interval is presented

10. Primary Outcome: Part B: Change From Baseline in Worst Knee Pain Intensity as Assessed by Numeric Rating Scale at Week 8
Description: Change from Baseline in worst knee pain intensity were assessed using NRS at Week 8. The pain NRS is an 11-point scale (ranging from 0-10) for self-reporting of average knee pain where 0 indicated no pain, and 10 indicated worst possible pain. The mean pain score prior to each visit was calculated as the average pain intensity in the 7 days prior to assessment visit. Participants were instructed to complete the pain NRS questionnaire at approximately the same time each day. A negative value change from baseline indicates an improvement. Baseline scores for each participant were assigned based on the first dosing visit.
Time Frame: Baseline (Day 1) and Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part B: Cohort 7: GSK3858279 | Part B: Placebo
Number analyzed (Participants) | 24 | 22
Scores on a scale | -2.89 (2.185) | -1.58 (2.057)
Statistical Analysis 1: Comparison: Part B: Cohort 7: GSK3858279 vs Part B: Placebo; Test type: Other — Bayesian Repeated Measures Model; Median Difference (Net) = -1.09, 95% CI 2-sided [-2.29 to 0.12], Standard Deviation 0.612 — Posterior median difference (GSK3858279 - Placebo) and 95% credible interval is presented

11. Secondary Outcome: Part A: Serum Concentrations of GSK3858279 Following a Single IV Dose
Time Frame: Up to 141 days
Reporting Status: Not Posted

12. Secondary Outcome: Part A: Serum Concentrations of GSK3858279 Following a Single SC Dose
Time Frame: Up to 141 days
Reporting Status: Not Posted

13. Secondary Outcome: Part B: Serum Concentration of GSK3858279 Following Repeat SC Dose
Time Frame: Up to 141 days
Reporting Status: Not Posted

14. Secondary Outcome: Part A: Area Under the Time-Concentration Curve (AUC) Over the Dosing Interval (0-tau) (AUC[0-tau]) Following a Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted, anticipated posting 2027-12

15. Secondary Outcome: Part A: AUC From Zero to Time t (0-t) (AUC[0-t]) Following a Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

16. Secondary Outcome: Part A: AUC From Zero to Infinity (0-infinity) (AUC[0-infinity]) Following a Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

17. Secondary Outcome: Part A: AUC(0-tau) Following a Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

18. Secondary Outcome: Part A: AUC From Zero to Time t (0-t) (AUC[0-t]) Following a Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

19. Secondary Outcome: Part A: AUC From Zero to Infinity (0-infinity) (AUC[0-infinity]) Following a Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

20. Secondary Outcome: Part B: AUC(0-tau) Following a Repeat SC Dose of GSK3858279
Time Frame: Baseline and Week 8
Reporting Status: Not Posted

21. Secondary Outcome: Part B: AUC(0-t) Following a Repeat SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

22. Secondary Outcome: Part B: AUC(0-infinity) Following a Repeat SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

23. Secondary Outcome: Part A: Maximum Concentration (Cmax) After a Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

24. Secondary Outcome: Part A: Maximum Concentration (Cmax) After a Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

25. Secondary Outcome: Part B: Cmax After Repeat SC Dose of GSK3858279
Time Frame: Baseline and Week 8
Reporting Status: Not Posted

26. Secondary Outcome: Part A: Half-life (t1/2) Following a Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

27. Secondary Outcome: Part A: Half-life (t1/2) Following a Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

28. Secondary Outcome: Part B: t1/2 Following a Repeat SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

29. Secondary Outcome: Part A: Clearance (CL) Following a Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

30. Secondary Outcome: Part A: Clearance (CL) Following a Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

31. Secondary Outcome: Part B: CL Following a Repeat SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

32. Secondary Outcome: Part A: Volume of Distribution at Steady State (Vss) Following a Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

33. Secondary Outcome: Part A: Volume of Distribution at Steady State (Vss) Following a Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

34. Secondary Outcome: Part B: Vss Following a Repeat SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

35. Secondary Outcome: Part A: Volume of Distribution (V) Following a Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

36. Secondary Outcome: Part A: Volume of Distribution (V) Following a Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

37. Secondary Outcome: Part B: Volume of Distribution (V) Following a Repeat SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

38. Secondary Outcome: Part A: Free Chemokine Ligand 17 (CCL17) Levels in Serum Following Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

39. Secondary Outcome: Part A: CCL17 Levels in Serum Following Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

40. Secondary Outcome: Part B: Free CCL17 Levels in Serum Following Repeat SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

41. Secondary Outcome: Part A: Total CCL17 Levels in Serum Following Single IV Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

42. Secondary Outcome: Part A: Total CCL17 Levels in Serum Following Single SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

43. Secondary Outcome: Part B: Total CCL17 Levels in Serum Following Repeat SC Dose of GSK3858279
Time Frame: Up to 141 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Part A and Part B: Up to 141 Days
Description: All-cause mortality, all non-serious treatment emergent Adverse events (TEAEs) and SAEs were collected. Safety population comprised of all randomized participants who received at least one dose of study treatment.
Arm/Group | Part A: Cohort 1: GSK3858279 | Part A: Cohort 2: GSK3858279 | Part A: Cohort 3: GSK3858279 | Part A: Cohort 4: GSK3858279 | Part A: Cohort 5: GSK3858279 | Part A: Cohort 6: GSK3858279 | Part A: Pooled Placebo | Part B: Cohort 7: GSK3858279 | Part B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 4/6 | 6/6 | 6/6 | 6/6 | 12/13 | 21/24 | 15/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1: GSK3858279 (N=6) | Part A: Cohort 2: GSK3858279 (N=6) | Part A: Cohort 3: GSK3858279 (N=6) | Part A: Cohort 4: GSK3858279 (N=6) | Part A: Cohort 5: GSK3858279 (N=6) | Part A: Cohort 6: GSK3858279 (N=6) | Part A: Pooled Placebo (N=13) | Part B: Cohort 7: GSK3858279 (N=24) | Part B: Placebo (N=24)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Administration site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sluggishness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 3 (4) | 3 (4) | 3 (3) | 2 (3)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (3) | 3 (5) | 2 (4) | 5 (11)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data has not been disclosed for pharmacokinetic parameters for this study as the development of the compound (GSK3858279) is still ongoing in another phase II study (NCT05838742) to fully understand the PK trends/parameters. We will disclose data for all pre-specified secondary PK parameters by 15-DEC-2027.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT03485365/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT03485365/SAP_001.pdf